CLINICAL TRIAL: NCT01683760
Title: Pharmacokinetic Study of Fluconazole in Premature Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han-Suk Kim, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FLU_PK; 12172_231 (Other Grant/Funding Number: Korea Food and Drug Administration)
Record Dates: First submitted 2012-09-09; First posted 2012-09-12 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Very Low Birth Weight Infant
Keywords: Fluconazole
MeSH Terms: interventions — Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Population PK (Experimental)
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Fluconazole — Prophylactic fluconazole administration in VLBW infants

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics of fluconazole which is used as prophylaxis of invasive fungal infection in premature infants.

ELIGIBILITY:
Inclusion Criteria:

* very low birth weight infant (birth weight < 1,500 g) who were admitted to the NICU before day 3 of life
* Informed consent from the parents

Exclusion Criteria:

* Major congenital anomaly
* Expired within 72 hours of life
* Liver failure (AST or ALT levels with three times the upper limit of the range of normal values or higher)
* Proven congenital or intrauterine fungal infection

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2012-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
drug level of fluconazole | 30min later, 10-12hr later, at routine lab with interval of 1week
  four times drug level after 3th dose

CONTACTS AND LOCATIONS:
Overall Officials: Han-Suk Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim YK, Lee J, Oh J, Rhee SJ, Shin SH, Yoon SH, Lee S, Kim HS, Yu KS. Population Pharmacokinetic Study of Prophylactic Fluconazole in Preterm Infants for Prevention of Invasive Candidiasis. Antimicrob Agents Chemother. 2019 May 24;63(6):e01960-18. doi: 10.1128/AAC.01960-18. Print 2019 Jun. PMID 30910892